CLINICAL TRIAL: NCT01877122
Title: Comparative Study of Safety and Efficacy of Heavyweight and Partially Absorbable Mesh in Inguinal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: MS1-1004
Record Dates: First submitted 2013-06-05; First posted 2013-06-13 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Hernia, Inguinal
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proflex® Mesh (Experimental): Device: Partially absorbable lightweight mesh Intervention: Mesh implantation
  Interventions: Device: Proflex® Mesh Mesh implantation
- Marlex® Mesh (Active Comparator): Device: Non-absorbable Heavyweight mesh Intervention: Mesh implantation
  Interventions: Device: Marlex® Mesh Implant

INTERVENTIONS:
Device: Proflex® Mesh Mesh implantation — Implantation of mesh in the incision of inguinal area
  Arms: Proflex® Mesh
Device: Marlex® Mesh Implant
  Arms: Marlex® Mesh

SUMMARY:
Proflex® Mesh (partially absorbable mesh, Korea) and Marlex® Mesh (heavyweight mesh) will be used for inguinal hernia repair to compare the safety and efficacy (pain score, quality of life)of two devices at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients >=20 years =<85 years old
2. Patients with Unilateral hernia
3. Patients without previous operations in lower part of abdomen
4. Patients capable to understand the explanation about purpose and method of the trial, and write an Informed Concent Form
5. Patients capable to participate during the period of the trial

Exclusion Criteria:

1. Previous hernia repair at the same site
2. Incarcerated hernia
3. Strangulated hernia
4. Patients to whom and open surgery cannot be indicated
5. Previous urological surgery
6. Immune incompetence of patient: AIDS, vesical fibrosis, etc.
7. Patients with AIHD or patients who take immunosuppressive drugs
8. Patients with liver disease (ASL, AST ≥ normal value by more than 3 times)
9. Patients with kidney disease (creatinine>2.0mg/dL)
10. Patients on anti-coagulants
11. Patients with severe systematic disease
12. Patients with malignant tumor
13. Patients with infection or with the predicted problem of surgery site healing
14. Participation in another clinical study within the last 30 days
15. Patients whose participation is considered inappropriate according to other except above mentioned clinical condition

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
pain score (10-point Visual Analogue Scale) | Day90 after operation

CONTACTS AND LOCATIONS:
Overall Officials: Taeil Son, M.D., Ph.D., Principal Investigator — Eulji Medical Center
Locations (1):
- Samyang Biopharmaceuticals, Seoul, South Korea